CLINICAL TRIAL: NCT05849415
Title: Correlation Between Periodontal Health, Psychological Stress and Mindfulness Awareness
Brief Title: Periodontal Health and Its Relationship With Psychological Stress
Status: Completed | Type: Observational
Sponsor: D'Albis Dental (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, DDS, Principal Investigator, University of Bari Aldo Moro
Other Study IDs: periodontology-stress
Record Dates: First submitted 2023-04-29; First posted 2023-05-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases; Stress; Mucositis; Periodontal
Keywords: Periodontal disease
MeSH Terms: conditions — Periodontal Diseases; Mucositis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Periodontal Screening and Recording, periodontal evaluation. — Periodontal probing for the evaluation of bleeding on probing and Periodontal Screening and Recording
  Other Names: Sheldon Cohen Perceived Stress Scale (PSS); Mindfulness Awareness Attention Scale (MAAS)

SUMMARY:
Studies suggest that chronic exposure to psychological stress can lead to oral health deterioration, alter the immune response, and possibly contribute to increased inflammation, which can impact the physiological healing of periodontal tissues.

People with psychophysiological stress disorders tend to acquire unhealthy habits, leading to less self-care, incorrect nutrition, smoking, alcohol consumption, and reduced physical activity.

This cross-sectional study aims to evaluate the correlation between periodontal health and psychological stress.

Patients between the ages of 35 and 70 will be recruited. Each patient must be visited and a periodontal assessment must be performed, recording the percentage of bleeding on probing and the Periodontal Screening and Recording (PSR). Subsequently, patients will be administered the Sheldon Cohen Perceived Stress Scale (PSS) and the Mindfulness Awareness Attention Scale (MAAS) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18

Exclusion Criteria:

* Pregnancy
* administration of antibiotics in the last 15 days prior to study entry or indications for antibiotic prophylaxis;
* orthodontic appliances
* immunological diseases or use of drugs that can affect oral tissues, (phenytoin, cyclosporine), nifedepine, chronic use of non-steroidal anti-inflammatory drugs);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: European people
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Periodontal health assessment | 4 month
  Periodontal Screening and Recording and percentage of bleeding on probing.
Sheldon Cohen Perceived Stress Scale (PSS) | 4 month
  The questionnaire consists of 10 questions regarding feelings and thoughts made during the last month. Possible answers have a value ranging from 0 to 4 based on the severity or frequency with which the person has thought in a certain way. For each question, the alternatives are as follows: 0 - never 1 - almost never 2 - sometimes 3 - fairly often 4 - very often. Therefore, the total score can range from 0 to 40. The range between 0 and 13 represents a perceived stress value that is either nonexistent or mild and well managed. The range between 14 and 26 represents a moderate stress value that can negatively affect physical and mental health. The range between 27 and 40 represents a perceived stress value that is severe and significantly compromises physical and mental health.
Mindfulness Awareness Attention Scale (MAAS) | 4 month
  Total score can range from 0 to 15. To measure the scale, one simply needs to calculate the average of the 15 responses.Higher scores reflect higher levels of disposition towards Mindfulness.

SECONDARY OUTCOMES:
relationship between periodontal health status and psychological tests | 4 month
  The results will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe D'Albis, Mola di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No